CLINICAL TRIAL: NCT02027064
Title: Interferon for the Intervention of Molecular Relapse in t (8; 21) AML After Allo-HSCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang, director of Peking University People's Hospital, institute of hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUPH IRB [2013](38)
Record Dates: First submitted 2014-01-02; First posted 2014-01-03 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Interferon-alpha

ARMS (1):
- interferon (Experimental)
  Interventions: Drug: Interferon-alpha

INTERVENTIONS:
Drug: Interferon-alpha

SUMMARY:
molecular relapse in t (8; 21) acute myeloid leukemia (AML) after allogeneic stem cell transplantation (allo-SCT) is still a problem even after donor lymphocyte infusion.

Interferon seemed to augment graft-versus-leukemia (GVL) effect in this part of patients.

the study is to evaluate the safety and efficacy of interferon for the intervention of molecular relapse in t (8; 21) acute myeloid leukemia (AML) after allogeneic stem cell transplantation (allo-SCT)

ELIGIBILITY:
Inclusion Criteria:

* high risk t (8; 21) AML
* molecular relapse after allo-SCT

Exclusion Criteria:

* active graft-versus-host disease
* uncontrolled severe infection
* organ function failure

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
relapse rate | participants will be followed for an expected average of 365 days
  number of participants with morphologic relapse at one year

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

REFERENCES:
- [Derived] Shen MZ, Zhang XH, Xu LP, Wang Y, Yan CH, Chen H, Chen YH, Han W, Wang FR, Wang JZ, Zhao XS, Qin YZ, Chang YJ, Liu KY, Huang XJ, Mo XD. Preemptive Interferon-alpha Therapy Could Protect Against Relapse and Improve Survival of Acute Myeloid Leukemia Patients After Allogeneic Hematopoietic Stem Cell Transplantation: Long-Term Results of Two Registry Studies. Front Immunol. 2022 Jan 28;13:757002. doi: 10.3389/fimmu.2022.757002. eCollection 2022. PMID 35154096
- [Derived] Mo XD, Wang Y, Zhang XH, Xu LP, Yan CH, Chen H, Chen YH, Qin YZ, Liu KY, Huang XJ. Interferon-alpha Is Effective for Treatment of Minimal Residual Disease in Patients with t(8;21) Acute Myeloid Leukemia After Allogeneic Hematopoietic Stem Cell Transplantation: Results of a Prospective Registry Study. Oncologist. 2018 Nov;23(11):1349-1357. doi: 10.1634/theoncologist.2017-0692. Epub 2018 Aug 3. PMID 30076280